## Effect of vitamin D supplementation on Graves' disease: The DAGMAR trial

| Patient Consent Form |
|--------------------------------------------|
| First approval January 25, 2013. |
| English translation August 16, 2022 |
| ClinicalTrials.gov Identifier: NCT02384668 |

## (S3) Informed consent for participation in a health science research project

| Title of research project: DAGMAR |
|---|
| Declaration from the study participant |
| I have received written and verbal information and I know enough about the purpose, method, |
| advantages and disadvantages to agree to participate |
| I know that <u>participation is voluntary</u> and that I can always withdraw my consent without losing my |
| current or future rights to treatment. |
| I consent to participate in the research project and have received a copy of this consent form and a copy of the written information about the project for my own use |
| Name of study subject: |
| Date:Signature: |
| Do you wish to be informed about the results of the research project and its potential implications for yourself? |
| Yes: No: |
| Statement from the person providing the information: |
| I declare that the study participant has received oral and written information about the research project. |
| In my opinion, sufficient information has been provided for a decision to be made regarding participation in the trial. |
| The name of the person who submitted the information: |
| Date:Signature: |
| Project identification: The Central Denmark Region Committees on Health Research Ethics, |

Standard declaration of consent prepared by the Scientific Ethics Committee System Denmark, December 2011

registration number 1-10-72-568-12